CLINICAL TRIAL: NCT02023372
Title: NuTech NuCel®: A Prospective, Efficacy Study of NuCel® in Patients Undergoing Fusion for One, Two or Three Level Degenerative Disease of the Lumbar Spine.
Brief Title: Efficacy Study of NuCel® in Patients Undergoing Fusion of the Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Carolina Neurosurgery & Spine Associates (Other); Wake Forest University Health Sciences (Other); Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2013-11-07
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Intervertebral Disc Disease; Intervertebral Disc Degeneration; Spondylosis; Spondylolisthesis; Spinal Stenosis
Keywords: NuCel; Lumbar Spine; Degenerative Disease; Efficacy; Fusion
MeSH Terms: conditions — Intervertebral disc disease; Intervertebral Disc Degeneration; Spondylosis; Spondylolisthesis; Spinal Stenosis | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NuCel with Autograft (Other): NuCel will be used with local autograft during surgical treatment of one, two or three level degenerative disease of the lumbar spine
  Interventions: Other: NuCel with Autograft

INTERVENTIONS:
Other: NuCel with Autograft — NuCel is a minimally manipulated allograft product derived from amniotic membrane along with cells from amniotic fluid. Local autograft is bone that comes from the patient's own vertebrae and surrounding bony structures.

SUMMARY:
The purpose of this study is to determine whether NuCel is effective in promoting spinal fusion in degenerative disease of the lumbar spine.

DETAILED DESCRIPTION:
The study is a prospective, single center clinical trial to establish the efficacy of NuCel, a minimally manipulated allograft tissue, for use in lumbar interbody and intertransverse fusion procedures. Subjects will undergo standard interbody fusion surgery as per the signed informed consent with NuCel and autograft bone. Patients will be evaluated postoperatively at 6 weeks, 3 months, 6 months, 1 year, and 2 years (if required).

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with degenerative disease of lumbar spine

Exclusion Criteria:

* Back pain due to injury
* Back pain that is caused by infection, cancer, lesions(growths) or bone disease such as osteoporosis
* Any terminal (will not recover from the disease) or autoimmune disease including but not limited to HIV infection, or rheumatoid arthritis
* Any other medical condition that might affect normal healing
* Less than 21 years of age
* More than three levels of fusion needed
* Recent history (within past 6 months) of any chemical or alcohol dependence
* Morbid obesity (Body Mass Index of more than 40)
* Currently a prisoner
* Currently experiencing a major mental illness
* Pregnancy at the time of enrollment
* Previously diagnosed with diseases of the bone such as osteoporosis, osteopenia or osteomalacia (softening of the bones). Patients with any of the risk factors for osteoporosis may have DEXA scans performed prior to study entry.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-12; Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Spinal Fusion | 12 months
  CT scan will be used to evaluate fusion of one, two, or three levels

SECONDARY OUTCOMES:
Change from baseline pain using Visual Analogue Scale (VAS) | 6 weeks, 3 months, 6 months, and 12 months
Change from baseline Oswestry Disability Index (Ver. 2.1) | 6 weeks, 3 months, 6 months, 12 months
X-ray to compare to baseline preoperative X-ray | 6 weeks, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Domagoj Coric, MD, Principal Investigator — Carolina Neurosurgery & Spine Associates
Locations (1):
- Carolina NeuroSurgery and Spine, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No